CLINICAL TRIAL: NCT03861169
Title: Prospective, Multi-Center, Single-Arm Post-Market Study of Use of the OMNI® Surgical System in Combination With Cataract Extraction in Open Angle Glaucoma
Brief Title: Study of OMNI System in OAG (GEMINI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sight Sciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06213
Record Dates: First submitted 2019-02-25; First posted 2019-03-04 (Actual); Results first posted 2024-08-14 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-07

CONDITIONS: Open Angle Glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle | interventions — Trabeculectomy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Viscoeleastic delivery & trabeculotomy (Experimental): Patients with open angle glaucoma and cataract
  Interventions: Device: Transluminal viscoelastic delivery and trabeculotomy

INTERVENTIONS:
Device: Transluminal viscoelastic delivery and trabeculotomy — Ab-interno transluminal viscoelastic delivery and trabeculotomy using OMNI Surgical System

SUMMARY:
This study will prospectively assess the clinical effect of ab-interno transluminal viscoelastic delivery and trabeculotomy performed using the OMNI Surgical System in combination with Cataract Extraction on intraocular pressure (IOP) and the use of IOP-lowering medications in patients with mild-moderate open angle glaucoma (OAG).

DETAILED DESCRIPTION:
This prospective, multicenter, single-arm, post-market clinical study will evaluate the impact of ab-interno transluminal viscoelastic delivery and trabeculotomy using OMNI Surgical System in conjunction with cataract surgery on IOP and the use of hypotensive medications in patients with mild to moderate open angle glaucoma.

ELIGIBILITY:
Inclusion Criteria:

Only one eye of each subject was eligible (the "study eye"), and all ocular criteria listed below applied to the study eye.

1. Male or female subjects, 22 years or older
2. Visually significant cataract
3. Diagnosed with mild to moderate open-angle glaucoma (e.g., primary open-angle glaucoma, pigmentary glaucoma, pseudoexfoliative glaucoma) as documented in subjects' medical record per ICD-10 guidelines
4. At screening, a medicated IOP ≤ 33 mmHg and on 1-4 IOP-lowering medications1 with a stable medication regimen for two months prior to screening visit
5. At baseline, unmedicated diurnal IOP 21-36 mmHg and IOP at least 3 mmHg higher than screening IOP
6. Scheduled for cataract extraction followed by ab- interno transluminal viscoelastic delivery and trabeculotomy using the OMNI Surgical System
7. Shaffer grade of ≥ 3 in all four quadrants
8. Potential of good best corrected visual acuity post cataract extraction, in the Investigator's judgment
9. Able and willing to comply with the protocol, including all follow-up visits.
10. Understood and signed the informed consent

Exclusion Criteria:

All criteria listed below applied to the study eye; both eyes of a single subject need not have been eligible for the study.

1. Any of the following prior treatments for glaucoma:

   * Laser trabeculoplasty ≤ 3 months prior to baseline
   * Implanted with iStent, CyPass, Xen, Express, glaucoma draining device/valve, or Hydrus Device
   * Prior canaloplasty, goniotomy, trabeculotomy, trabeculectomy, ECP or CPC
2. Normal tension glaucoma
3. Acute angle closure, traumatic, congenital, malignant, uveitic or neovascular glaucoma
4. Severe glaucoma as documented in subjects' medical record per ICD-10 guidelines
5. Use of oral hypotensive medication treatment for glaucoma
6. In the Investigator's judgement, predisposed to significant risk because of washout of ocular hypotensive medications
7. Ocular pathology or medical condition which, in the Investigator's judgment, would either place the subject at increased risk of complications, contraindicate surgery, place the subject at risk of significant vision loss during the study period (e.g., wet AMD, corneal edema, Fuch's dystrophy, etc.), or interfere with compliance to elements of the study protocol (e.g., returning to Investigator's office for follow-up visits)
8. Participation (≤ 30 days prior to baseline) in an interventional trial which could have a potential effect on the study outcome, as determined by the study investigator
9. Women of childbearing potential if they are currently pregnant or intend to become pregnant during the study period; are breast-feeding; or are not in agreement to use adequate birth control methods to prevent pregnancy throughout the study

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 209 (Actual)
Dates: Start 2019-03-11 (Actual); Primary Completion 2021-05-04 (Actual); Study Completion 2021-05-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jaime Dickerson, PhD, Study Director — Sight Sciences
Locations (15):
- United States (15):
  - Eye Center South, Dothan, Alabama
  - Barnet Delaney Perkins Eye Center, Lake Havasu City, Arizona
  - Vold Vision, Fayetteville, Arkansas
  - Your Eye Specialists, Weston, Florida
  - Omni Eye Services, Atlanta, Georgia
  - Eye Physicians and Surgeons, LLP, Iowa City, Iowa
  - Grene Vision Group, Wichita, Kansas
  - Vance Thompson Vision - MT, Bozeman, Montana
  - Vance Thompson Vision - NE, Omaha, Nebraska
  - Vance Thompson Vision - ND, West Fargo, North Dakota
  - Oklahoma Eye Surgeons, Oklahoma City, Oklahoma
  - Northern Ophthalmics, Jenkintown, Pennsylvania
  - El Paso Eye Surgeons, El Paso, Texas
  - Ophthalmology Associates, Fort Worth, Texas
  - Eye Centers of Racine and Kenosha, Kenosha, Wisconsin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- OMNI® Surgical System: Cataract extraction followed by ab-interno transluminal viscoelastic delivery and trabeculotomy using the OMNI Surgical System
Period: Overall Study
Arm/Group | OMNI® Surgical System
Started | 209
Completed | 149
Not Completed | 60

BASELINE CHARACTERISTICS:
Groups:
- OMNI® Surgical System: Eligible subjects had cataract and mild-moderate OAG with intraocular pressure (IOP) ≤33 mmHg on 1 to 4 hypotensive medications at Screening and Cataract extraction followed by ab-interno transluminal viscoelastic delivery and trabeculotomy using the OMNI Surgical System
Arm/Group | OMNI® Surgical System
Number analyzed (Participants) | 149
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: Across three study populations (Safety/ITT, mITT, PP)
  Years
    ITT/Safety Population | 68.3 (8.5)
    mITT: number analyzed (Participants) | 141
    mITT | 68.6 (8.3)
    Per Protocol Population: number analyzed (Participants) | 120
    Per Protocol Population | 68.8 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Across three study populations (Safety/ITT, mITT, PP)
  Participants
    ITT/Safety Population: Female | 89
    ITT/Safety Population: Male | 60
    mITT: number analyzed (Participants) | 141
    mITT: Female | 85
    mITT: Male | 56
    Per Protocol Population: number analyzed (Participants) | 120
    Per Protocol Population: Female | 73
    Per Protocol Population: Male | 47
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Across three study populations (Safety/ITT, mITT, PP)
  Participants
    ITT/Safety Population: Hispanic or Latino | 41
    ITT/Safety Population: Not Hispanic or Latino | 108
    ITT/Safety Population: Unknown or Not Reported | 0
    mITT: number analyzed (Participants) | 141
    mITT: Hispanic or Latino | 38
    mITT: Not Hispanic or Latino | 103
    mITT: Unknown or Not Reported | 0
    Per Protocol: number analyzed (Participants) | 120
    Per Protocol: Hispanic or Latino | 30
    Per Protocol: Not Hispanic or Latino | 90
    Per Protocol: Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Across three study populations (Safety/ITT, mITT, PP)
  Participants
    ITT/Safety Population: American Indian or Alaska Native | 1
    ITT/Safety Population: Asian | 2
    ITT/Safety Population: Native Hawaiian or Other Pacific Islander | 0
    ITT/Safety Population: Black or African American | 24
    ITT/Safety Population: White | 122
    ITT/Safety Population: More than one race | 0
    ITT/Safety Population: Unknown or Not Reported | 0
    mITT: number analyzed (Participants) | 141
    mITT: American Indian or Alaska Native | 1
    mITT: Asian | 2
    mITT: Native Hawaiian or Other Pacific Islander | 0
    mITT: Black or African American | 23
    mITT: White | 115
    mITT: More than one race | 0
    mITT: Unknown or Not Reported | 0
    Per Protocol: number analyzed (Participants) | 120
    Per Protocol: American Indian or Alaska Native | 1
    Per Protocol: Asian | 0
    Per Protocol: Native Hawaiian or Other Pacific Islander | 0
    Per Protocol: Black or African American | 19
    Per Protocol: White | 100
    Per Protocol: More than one race | 0
    Per Protocol: Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 149
Study Eye [Count of Participants; unit: Participants] — Population: Across three study populations (Safety/ITT, mITT, PP)
  Participants
    ITT/Safety Population: OD | 74
    ITT/Safety Population: OS | 75
    mITT: number analyzed (Participants) | 141
    mITT: OD | 70
    mITT: OS | 71
    Per Protocol Population: number analyzed (Participants) | 120
    Per Protocol Population: OD | 58
    Per Protocol Population: OS | 62
Glaucoma Status [Count of Participants; unit: Participants] — Population: Across three study populations (Safety/ITT, mITT, PP)
  Participants
    ITT/Safety Population: Primary Open Angle Glaucoma | 139
    ITT/Safety Population: Pigmentary | 1
    ITT/Safety Population: Pseudoexfoliative | 9
    mITT: number analyzed (Participants) | 141
    mITT: Primary Open Angle Glaucoma | 131
    mITT: Pigmentary | 1
    mITT: Pseudoexfoliative | 9
    Per Protocol Population: number analyzed (Participants) | 120
    Per Protocol Population: Primary Open Angle Glaucoma | 113
    Per Protocol Population: Pigmentary | 1
    Per Protocol Population: Pseudoexfoliative | 6

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Unmedicated Diurnal IOP
Description: Change in mean unmedicated diurnal IOP from baseline to 12 months
Time Frame: 12 months
Population: The Per Protocol (PP) analysis population was a subset of the mITT population and included all subjects who were on least one ocular hypotensive medication at screening and had uneventful cataract extraction followed by ab-interno transluminal viscoelastic delivery and trabeculotomy, 12 month IOP and medication data, and had no clinically significant protocol deviations.
Measure: Mean (Standard Deviation); unit: mm Hg
Groups:
- Per Protocol Population: Primary inference was based on the PP population.
Arm/Group | Per Protocol Population
Number analyzed (Participants) | 120
mm Hg | 7.98 (4.21)

2. Primary Outcome: Change in Mean Number of IOP-Lowering Medications
Description: Reduction in mean number of IOP-lowering medications from screening to 12 months
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: medications
Arm/Group | Per Protocol Population
Number analyzed (Participants) | 120
medications | 1.43 (1.14)

3. Secondary Outcome: Percent of Eyes With a ≥20% Reduction in Unmedicated DIOP
Description: First Secondary Effectiveness endpoint/Percent of eyes with a ≥20% reduction in unmedicated DIOP at 12 months
Time Frame: 12 months
Measure: Number; unit: percentage of eyes
Groups:
- Per Protocol Population: Based on Per Protocol population.
- mITT: Based on mITT population.
Arm/Group | Per Protocol Population | mITT
Number analyzed (Participants) | 120 | 141
percentage of eyes | 84.2 | 75.9

4. Secondary Outcome: Percent of Eyes With Unmedicated Diurnal IOP Between 6 and 18 mmHg Inclusive at 12 Months
Description: Second Secondary Effectiveness Endpoint: Unmedicated DIOP ≥ 6 mmHg and ≤ 18 mmHg at 12 Months/Percent of eyes with unmedicated DIOP between 6 and 18 mmHg inclusive at 12 months
Time Frame: 12 months
Measure: Number; unit: percentage of eyes
Arm/Group | Per Protocol Population | mITT
Number analyzed (Participants) | 120 | 141
percentage of eyes | 77.5 | 70.9

ADVERSE EVENTS:
Time Frame: 12 Months
Groups:
- iTT/Safety: The ITT/Safety population, defined as all enrolled and treated subjects regardless of whether or not they had a protocol deviation, comprised 149 subjects. All safety evaluations were performed on this population.
Arm/Group | iTT/Safety
All-Cause Mortality (participants affected / at risk) | 34/149
Serious Adverse Events (participants affected / at risk) | 2/149
Other Adverse Events (participants affected / at risk) | 34/149
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | iTT/Safety (N=149)
Torn rotator cuff subsequent to fainting (Unrelated) (Musculoskeletal and connective tissue disorders) | 1 (1)
Bradycardia (Unrelated) (Cardiac disorders) | 1 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | iTT/Safety (N=149)
Posterior capsular tear (Eye disorders) | 2 (2)
Loss of 2 lines or more BCVA (10 or more ETDRS letters) at or after 3 months postoperative (Eye disorders) | 2 (2)
Chronic anterior uveitis (Eye disorders) | 2 (3) — Inflammation of grade 1+ or worse persisting for more than 3 months post-operatively or that recurs less than three months after discontinuing treatment
Layered hyphema greater than or equal to 1mm (Eye disorders) | 9 (9)
Peripheral Anterior Synechiae >1 clock hour (Eye disorders) | 2 (2)
Vitreous hemorrhage (Eye disorders) | 1 (1)
Clinically significant cystoid macular edema (Eye disorders) | 1 (1)
Increase in C/D ratio of > 0.3 units compared to baseline on slit lamp exam (Eye disorders) | 2 (2)
IOP increase requiring management with systemic medication at greater than or equal to 1 month visit (Eye disorders) | 2 (2)
IOP increase greater than or equal to 10 mmHg above baseline IOP at greater than or equal to 1M (Eye disorders) | 3 (3)
Blepharitis (Eye disorders) | 3 (3)
Cystoid macular edema (CME) (Eye disorders) | 2 (2)
Dry Eye (Eye disorders) | 1 (1)
Guttae (Eye disorders) | 1 (1)
Hordeolum (Eye disorders) | 1 (1)
Iritis (Eye disorders) | 2 (2)
Microhyphema (Eye disorders) | 2 (2)
Ocular migraine (Eye disorders) | 1 (1)
Posterior capsular opacification (PCO) (Eye disorders) | 5 (5)
Superficial punctate keratitis (SPK) (Eye disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-01): https://cdn.clinicaltrials.gov/large-docs/69/NCT03861169/Prot_SAP_001.pdf